CLINICAL TRIAL: NCT06611943
Title: DietCoach: Development and Dietitian Evaluation of a Digital Dietary Counseling Platform
Acronym: DietCoach
Status: Recruiting | Type: Observational
Sponsor: University of St.Gallen (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Wu Jing, Ph.D. Candidate and Project Leader, University of St.Gallen
Other Study IDs: UStGallen
Record Dates: First submitted 2024-09-09; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Dietary Habits; Food Habits; Nutrition, Healthy; Diet, Healthy
Keywords: Digital dietary counseling; Food purchase data; Dietitian interface; eHealth; Human-Computer Interaction
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Low patient food shopping coverage: In this group, participants need to give at least one dietary recommendation to a patient whose loyalty card(s) cover(s) a low percentage of food purchases.
  Interventions: Behavioral: DietCoach
- Medium patient food shopping coverage: In this group, participants need to give at least one dietary recommendation to a patient whose loyalty card(s) cover(s) a medium percentage of their food purchases.
  Interventions: Behavioral: DietCoach
- High patient food shopping coverage: In this group, participants need to give to at least one dietary recommendation to a patient whose loyalty card(s) cover(s) a high percentage of food purchases.
  Interventions: Behavioral: DietCoach

INTERVENTIONS:
Behavioral: DietCoach — Participants are invited to give at least one dietary recommendation to a patient's food purchase data using the DietCoach platform.

SUMMARY:
The DietCoach study aims to investigate the requirements of a digital dietary counseling platform, and evaluate the dietitian acceptance and usability of the DietCoach platform, which was developed based on the collected requirements. Additionally, the study examines how different levels of patient food purchase data availability affect these factors. The DietCoach platform automatically tracks historic and up-to-date patient food purchase data on loyalty cards and provides nutritional analysis, assisting dietitians in the dietary counseling process. The key research questions (RQ) are:

1. What are the requirements of a digital dietary counseling system based on food purchase data?
2. What is acceptance and usability of the DietCoach platform evaluated by dietitians?
3. How does the availability of patient food purchase data influence the acceptance and perceived usability of the DietCoach platform by dietitians?

Dietitians from several cantonal hospitals in the German-speaking area of Switzerland are invited to participate in the study. To answer RQ1, we conduct a workshop and a survey with dietitians to derive key requirements on dietary counseling systems. To answer RQ2 and RQ3, we use a cross-sectional, mixed-methods, between-subjects study design.

Researchers will evaluate and compare the acceptance and usability of DietCoach in 3 different conditions (3 patients that had different, i.e., high, medium and low, food purchase data availability). Each participant is assigned to the data of one patient. Participants are required to:

1. use the DietCoach platform to provide at least one dietary recommendation to patient food purchase data in two separate sessions.
2. provide quantitative and qualitative feedback about the acceptance and usability of the DietCoach platform.

DETAILED DESCRIPTION:
The DietCoach study aims to investigate the requirements of a digital dietary counseling platform, and evaluate the dietitian acceptance and usability of the DietCoach platform, which was developed based on the collected requirements. Additionally, the study examines how different levels of patient food purchase data availability affect these factors. The DietCoach platform automatically tracks historic and up-to-date patient food purchases on loyalty cards and provides nutritional analysis.

Dietitians from several cantonal hospitals in the German-speaking area of Switzerland are invited to participate. To collect the key requirements of a digital dietary counseling platform based on food purchase data, we conduct a workshop and a survey, using guiding questions designed based on our research over the last years. To understand the acceptance and usability of DietCoach and how food purchase data availability influences these factors, we use a cross-sectional, mixed-methods, between-subjects study design. Each participant is assigned to the data of one patient. Participants need to:

1. use the DietCoach platform to provide at least one dietary recommendation to patient food purchase data in two separate sessions.
2. provide quantitative and qualitative feedback about the acceptance and usability of the DietCoach platform.

The DietCoach usability study includes three conditions (data from three patients), defined by High, Medium, and Low levels of patient food purchase data availability. Data availability is determined by the number of baskets/items (from the major Swiss retail chain) per person in a patient household. Participants are randomly assigned to the data of one patient.

In both the initial and follow-up sessions, participants need to provide at least one dietary recommendation based on the patient's health status and food purchase data over 8 weeks. The food purchase data in the follow-up session covers the 8 weeks immediately following those considered in the initial session. After completing the assigned tasks on the platform, participants are asked to complete a survey assessing their acceptance of and the usability of the DietCoach platform.

ELIGIBILITY:
Inclusion Criteria:

* Dietitians in Switzerland
* German-speaking (the platform is in German, a main language in Switzerland)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study aims to include all dietitians in Switzerland as potential participants. However, since recruitment will be conducted through contacting the nutritional departments of cantonal hospitals in the German-speaking area, the participant pool is expected to consist primarily of dietitians from several cantonal hospitals located in the German-speaking region of Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Key requirements of a digital dietary counseling system based on food purchase data | Immediately after the DietCoach intervention
  The key requirements for a digital dietary counseling system based on food purchase data will be identified through the dietitian workshop and the dietitian survey. They primarily focus on:
  1. food purchase data availability: number of baskets/items per person in a patient household, and the duration of data availability.
  2. use cases: percentage of participants identifying critical use cases (e.g., recommending alternative food products).
  3. product information: most important product information (e.g., energy, sugar) identified by dietitians for a dietary counseling system.
  All outcomes will be quantified using a 5-point Likert scale (from 1 very low importance to 5 very high importance), according to participant responses. Participants are additionally allowed to add more suggestions/recommendation/comments using free text.
Acceptance of the DietCoach platform | Immediately after the DietCoach intervention
  Evaluated by the modified Unified Theory of Acceptance and Use of Technology (UTAUT2) constructs. The constructs include performance expectancy, effort expectancy, facilitating conditions, hedonic motivation and behavioral intention.
  The construct levels can be indicated by the average score on a 7-point Likert scale.
Usability of the DietCoach platform | Immediately after the DietCoach intervention
  Measured by the average System Usability Scale (SUS) score, ranging from 0 to 100. The higher the SUS score, the better the usability

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wu, M.Sc., Principal Investigator — University of St.Gallen
Locations (1):
- University of St.Gallen, Sankt Gallen, St.Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
We plan to publish anonymized partial food purchase data of the selected patients, and the corresponding dietary recommendations from the DietCoach study participants (dietitians)
  1. The data will be published in an anonymized form.
  2. Only purchase records that can be identified by our food composition database and belong to relevant food categories will be published.
Supporting Information: SAP
Time Frame: The data will become available in 2024/2025, published as supplementary materials to the corresponding paper to ensure the result reproducibility. It will be available until participants request to delete their data. Published aggregated results could not be withdrawn retrospectively.